CLINICAL TRIAL: NCT02779673
Title: Investigation of the Effectiveness of Plant Stanols as Ester on Change in Blood Cholesterol Level in Korean Adult
Brief Title: The Effectiveness of Plant Stanols as Ester on Change in Blood Cholesterol Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LF_cholesterol
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: LDL-cholesterol Level 130-159mg/dL
MeSH Terms: interventions — Esters; Sitosterols

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Test group (Experimental): Subjects randomized to the test group consumed yoghurt drink containing 3.4g plant stanol as ester for 1 per day for a period of 4 weeks.
  Interventions: Other: Yoghurt drink containing plant stanol as esters
- Placebo group (Placebo Comparator): Subjects randomized to the placebo group consumed yoghurt drink without plant stanol as ester for 1 per day for a period of 4 weeks.
  Interventions: Other: Yoghurt drink without plant stanol as esters

INTERVENTIONS:
Other: Yoghurt drink containing plant stanol as esters
  Arms: Test group
Other: Yoghurt drink without plant stanol as esters
  Arms: Placebo group

SUMMARY:
The purpose of randomized, double-blind, placebo-controlled study was to determine whether yoghurt drink containing 2g plant stanols (3.4g as plant stanol esters) is effective in the control of blood cholesterol level in subjects with LDL-cholesterol level 130-159mg/dL.

DETAILED DESCRIPTION:
The objective of clinical trial was to evaluate the effect of yoghurt drink containing 2g plant stanols (3.4g as plant stanol esters) on blood cholesterol level. A randomized, double-blinded, placebo-controlled study was conducted on subjects with LDL-cholesterol level 130-159mg/dL. The subjects were randomly assigned to either a group ingesting yoghurt drink containing 2g plant stanols (3.4g as plant stanol esters) or a placebo group (yoghurt drink without plant stanols) for 4-week. The investigators assessed blood cholesterol level.

ELIGIBILITY:
Inclusion Criteria:

• LDL-cholesterol level 130-159mg/dL (not taking cholesterol-lowering medications)

Exclusion Criteria:

* taking any medications (including anti-hypertensive, lipid lowering, anti-platelets, and anti-diabetic drugs)
* history of serious cardiovascular, pulmonary, gastrointestinal, hepatic, renal and/or haematological disease
* history or presence of cancer
* history of a psychiatric disorder and/or drug or alcohol abuse or dependency;
* having a known intolerance to gluten or lactose
* having a known allergy to any ingredient in the investigational product
* women who are pregnant or desire to become pregnant during the study period or within 3 months of giving birth or breast feeding or within 3 months of cessation of breast feeding
* having any other medical condition which, in the opinion of the investigator, could interfere with participation in the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline LDL-cholesterol at 4-week | at baseline and 4-week follow-up
Change from baseline total cholesterol at 4-week | at baseline and 4-week follow-up
Change from baseline non-HDL-cholesterol at 4-week | at baseline and 4-week follow-up

SECONDARY OUTCOMES:
Change from baseline triglyceride at 4-week | at baseline and 4-week follow-up
Change from baseline HDL-cholesterol at 4-week | at baseline and 4-week follow-up
Change from baseline Apolipoprotein A1 at 4-week | at baseline and 4-week follow-up
Change from baseline Apolipoprotein B at 4-week | at baseline and 4-week follow-up